CLINICAL TRIAL: NCT06136403
Title: A 44-week Monocentric Open Study Assessing the Efficacy and Safety of Deucravacitinib in Adults With Inflammatory Genodermatoses
Acronym: GENEPID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-PP-20; 2022-502879-32-00 (Other: CTIS)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Epidermolysis Bullosa Simplex; Ichthyosis; Genodermatosis; Inflammatory Congenital Ichthyoses
Keywords: deucravacitinib
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Ichthyosis; Skin Diseases, Genetic | interventions — deucravacitinib

STUDY DESIGN:
Intervention Model Description: challenge dechalenge rechalenge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- deucravacitinib treatment (Experimental): challenge-dechallenge -rechallenge design
  Interventions: Drug: deucravacitinib

INTERVENTIONS:
Drug: deucravacitinib — treatment by deucravacitinib in two phases of challenge

SUMMARY:
The goal of this clinical trial is to learn about deucravacitinib treatment in adults with inflammatory epidermal genodermatoses . The main question it aims to answer are: describe efficacity and safety of this treatment.

Participants will take treatments and have to use bullets during the study period.

DETAILED DESCRIPTION:
The patient will have 8 visits After Confirmation of inclusion criteria and no exclusion criteria, the study will be explain to the patient after signing the inform consent and be included in the study Treatment Period (Period 1); challenge period This period will be the first treatment period that will occur from 16 weeks. During this period the patient will see the doctor at the hospital, he will perform the study procedures The second period : dechallenge (period 2): All patients stop their treatment for 12 weeks.

The second treatment period - rechallenge (period 3) the patient will take the treatment for a second 16 weeks period At week 44 - End of study

At each visit:

The investigator at each visit compliance to the treatment and adverse events, Measure vital signs and perform clinical examination.

The patient will assess the different questionnaires, for the study and have blood sample

ELIGIBILITY:
Inclusion Criteria:

* Subject has congenital skin fragility with skin and/or mucosal blisters, a clinical phenotype of EBS-sev and a laboratory confirmed diagnosis of EBS by KRT5 and/or 14 mutation (autosomal only) OR a clinical phenotype of inflammatory ichthyosis (IC) including keratinopathic ichthyosis due to KRT1/10 mutation, ECI with identified genetic mutations (TGM5, NIPAL4, ABCA12, etc…).
* Subject has at least a mean daily number of 4 new blisters (EBS-sev) OR an ISS > 50/128.

  * Subject agrees not to use any topical therapies other than the investigator approved.

Exclusion Criteria:

* Subjects with another form of ICI ie Netherton syndrome, Kid syndrome etc.
* Infectious/Immune-related Exclusions
* Medical History and Concurrent Diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of deucravacitinib | week 44
  number of new blister conting every day

SECONDARY OUTCOMES:
Safety of deucravacitinib treatment | week 44
  record of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chiaverini, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice, Nice, CHU de NICE
  - APHP St Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No